CLINICAL TRIAL: NCT01222351
Title: BAY 94-9172 PET/CT in Cognitively Normal Older Adults, Older Adults With Mild Cognitive Impairment, and Older Adults With Alzheimer's Disease
Brief Title: Measuring Brain Amyloid Plaque Load in Older Adults Using BAY 94-9172
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Bayer (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yaakov Stern, Professor of Neuropsychology, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6045/7130R (Bayer); IND 78868 (Other: U.S. Food and Drug Administration); R01AG037212-01 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Late Onset Alzheimer Disease
Keywords: Alzheimer's disease; Positron emission tomography; Biomarker; Brain amyloid plaque load
MeSH Terms: conditions — Alzheimer Disease | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAY 94-9172 (Experimental): BAY 94-9172 PET/CT
  Interventions: Drug: BAY 94-9172 (Florbetaben)

INTERVENTIONS:
Drug: BAY 94-9172 (Florbetaben) — Measure of brain amyloid load using BAY 94-9172 PET/CT
  Other Names: Florbetaben; Bay 91-9172

SUMMARY:
The overall goal of this project is to establish and validate biomarkers associated with the risk and progression of late onset Alzheimer's disease, mild cognitive impairment and cognitive decline. The investigators will use baseline and longitudinal measurements of plasma amyloid beta-40 and amyloid beta-42 to investigate the risk of developing mild cognitive impairment and late onset Alzheimer's disease, as well as the rates of cognitive decline and Alzheimer's disease progression. The driving hypothesis of the study is that amyloid beta in the brain as measured by positron emission tomography positivity is associated with the onset of cognitive decline associated with late onset Alzheimer's disease.

DETAILED DESCRIPTION:
This project is a sub-study of the Washington Heights-Inwood Community Aging Project, which is a multidisciplinary, epidemiological study of Alzheimer's disease and related neurodegenerative disorders. We will obtain positron emission tomography scans and simultaneous x-ray computed tomography scans using Florbetaben from Bayer on a selection of ongoing participants who will be selected on the basis of change in plasma levels of amyloid beta over time. Approximately 200 participants will receive scans beginning in 2009 and in the 2010-2012 assessment wave and then again in a 2014-2015 assessment wave. Our intention is to examine whether uptake of Florbetaben in the brain is associated with decline in cognition over the 10 years prior to the PET scan.

ELIGIBILITY:
Inclusion Criteria:

* Current Washington Heights-Inwood Community Aging Project (WHICAP) participant Age 65 or older Residing in the community of Washington-Heights/Inwood/Hamilton Heights
* Is able to provide informed consent, understand the information provided on the purpose and conduct of the trial and exhibits adequate visual, auditory and communication capabilities to enable compliance with study procedures. This includes performing the psychometric testing and being able to lie down flat in the Positron Emission Tomography (PET) scanner
* Possesses a general health that permits adequate compliance with all study procedures.
* Informed consent has been signed and dated (with time) by the subject and/or the subject's caregiver (for probable Alzheimer's Disease (AD) patients)

Exclusion Criteria:

* Has any contraindication to PET, such as claustrophobia, or inability to lie flat for half an hour as determined by the onsite radiologist performing the scan
* Current, past, or anticipated exposure to radiation, which may include being badged for radiation exposure in the workplace or participation in nuclear medicine procedures, including research protocols in the last year
* Significant active physical illness particularly those that may affect the brain including blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure or chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, low hemoglobin and malignancy
* Scheduled for surgery and/or another invasive procedure within the time period of up to 24 hours following scan
* Allergic to the tracer or any of its constituents and/or has a history of severe allergic reactions to drugs or allergens (e.g. patients with allergic asthma)
* Critically ill and/or medically unstable and whose clinical course within the observation period is unpredictable, e.g. participants with 14 days of myocardial infarction or stroke, unstable participants with previous surgery (within 7 days), participants with advanced heart insufficiency (New York Heart Association (NYHA) stage IV), or participants with acute renal failure.
* Has received any contrast material (X-ray, Magnetic Resonance Imaging (MRI)), or radiopharmaceuticals within 48 hours prior to the application of the Investigational Medicinal Product (IMP) or for whom application of such a substance is planned for 24 hours following IMP administration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2014-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mayeux, BS, MD, MSc, Principal Investigator — Columbia University; Yaakov Stern, BA, PhD, Study Chair — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Cosentino SA, Stern Y, Sokolov E, Scarmeas N, Manly JJ, Tang MX, Schupf N, Mayeux RP. Plasma ss-amyloid and cognitive decline. Arch Neurol. 2010 Dec;67(12):1485-90. doi: 10.1001/archneurol.2010.189. Epub 2010 Aug 9. PMID 20697031
- [Background] Forsberg A, Almkvist O, Engler H, Wall A, Langstrom B, Nordberg A. High PIB retention in Alzheimer's disease is an early event with complex relationship with CSF biomarkers and functional parameters. Curr Alzheimer Res. 2010 Feb;7(1):56-66. doi: 10.2174/156720510790274446. PMID 20205671
- [Result] Gu Y, Razlighi QR, Zahodne LB, Janicki SC, Ichise M, Manly JJ, Devanand DP, Brickman AM, Schupf N, Mayeux R, Stern Y. Brain Amyloid Deposition and Longitudinal Cognitive Decline in Nondemented Older Subjects: Results from a Multi-Ethnic Population. PLoS One. 2015 Jul 29;10(7):e0123743. doi: 10.1371/journal.pone.0123743. eCollection 2015. PMID 26221954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BAY 94-9172
Started | 160
Completed | 160
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BAY 94-9172
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 67
  White | 58
  More than one race | 12
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  United States | 160

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Cognitive Change Over Time and Amyloid (Aβ) Deposition
Description: We used PET imaging to measure presence of amyloid. The outcomes are cognitive z-scores, which had mean of zero and SD of 1, with no units. There are four cognitive domains (language, memory, processing speed, and visuospatial ability). Individual neuropsychological test Z-scores within each domain were averaged to get the mean domain z-scores. Finally, the four cognitive domain-specific Z-scores were then averaged into a global cognitive Z-score. A larger Z-score represents better cognitive performance.
  Latent growth curve model was used to test for the association between Aβ and cognitive change over time. The Beta weight is a coefficient from the model that indicates the difference in cognitive change between people with and without amyloid. A positive Beta weight indicates that Aβ deposition is associated with less decline in cognitive scores, a negative Beta weight indicates greater decline. The Beta weight is unitless, and it does not have a range.
Time Frame: up to 3 years and 10 months
Population: In this analysis we evaluated whether the presence of amyloid was related to previous decline in cognition in 116 subjects. Mean cognition summarized performance on several cognitive tests. were analyzed. Global amyloid burden was rated with a visual rating by 2 trained clinicians.
Measure: Count of Participants; unit: Participants
Groups:
- BAY 94-9172: We used BAY 94-9172 (Florbetaben) to measure the presence of of brain amyloid.
Arm/Group | BAY 94-9172
Number analyzed (Participants) | 116
Participants
  Participant with positive amyloid reading | 41
  Participant without positive amyloid reading | 75
Statistical Analysis 1: Comparison: BAY 94-9172; Test type: Equivalence — The null hypothesis was that there is no difference in the rate of cognitive decline between participants with and without amyloid; p = 0.02, latent growth curve model; Latent growth curve models tested cognitive decline rate by amyloid status; Slope = -0.034 — B weights were the estimates for the association between Aβ and cognitive change

ADVERSE EVENTS:
Arm/Group | BAY 94-9172
All-Cause Mortality (participants affected / at risk) | 0/160
Serious Adverse Events (participants affected / at risk) | 0/160
Other Adverse Events (participants affected / at risk) | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes